CLINICAL TRIAL: NCT07173595
Title: A Phase I Clinical Study to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of QLS2309 Injection in Patients With CD70+ Relapsed/Refractory Hematologic Malignancies
Brief Title: A Phase I Study of QLS2309 Injection in Patients With CD70+ Relapsed/Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS2309-101
Record Dates: First submitted 2025-09-05; First posted 2025-09-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Hematologic Malignancies
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS2309 (Experimental)
  Interventions: Drug: QLS2309

INTERVENTIONS:
Drug: QLS2309 — initial dose - MTD; QW; intravenous infusion

SUMMARY:
This is a single-arm, open-label, multicenter, dose-escalation, dose-expansion and efficacy-expansion phase I clinical study to evaluate the tolerability, safety, pharmacokinetics and preliminary antitumor activity of QLS2309 injection in patients with CD70+ relapsed/refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily participated and signed a written informed consent form
* Age ≥ 18 years, male or female
* ECOG performance status of 0-2
* Expected life-expectancy ≥ 3 months
* CD70+ relapsed/refractory hematologic malignancies
* Adequate organ function prior to QLS2309 administration
* Female patients with fertility must agree to the use of effective contraceptive methods during the study period and within 35 days of discontinuation of the trial drug.
* Male patients whose sexual partners are women of childbearing age must agree to use condoms during the study period and within 35 days of discontinuation of the trial drug during sexual intercourse.

Exclusion Criteria:

* Prior treatment with CD70-related antibodies, antibody-conjugated drugs (ADCs) or cell therapy products
* Symptomatic central nervous system (CNS) involvement, leptomeningeal metastasis or spinal cord compression caused by metastasis
* An active autoimmune diseases or known history of ≥ grade 3 irAE due to prior immunotherapy
* Known history of other active malignant tumor within 3 years
* Known history of chemotherapy, biological therapy, endocrine therapy, immunotherapy, monoclonal antibodies, etc. within 4 weeks
* Known history of active hepatitis B/C infection, HIV infection, Treponema pallidum infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 28 days
  To evaluate the safety and tolerability of QLS2309
Recommended Phase Ib Dose (RPIbD) | up to 2 years
  The Safety Monitoring Committee (SMC) will select RP1bD based on the safety, tolerability, PK parameters, pharmacodynamics, preliminary effectiveness and other data of subjects in different dose groups

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China